CLINICAL TRIAL: NCT04960137
Title: Non-randomized Controlled Study of Shoulder Dislocations Treated With Button Plates and Non-absorbable Suture Anchor
Brief Title: Shoulder Dislocations Treated With Button Plates and Non-absorbable Suture Anchor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Hunan People's Hospital (Unknown); The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D2016052
Record Dates: First submitted 2021-07-04; First posted 2021-07-13 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Shoulder Dislocation
Keywords: button; non-absorbable suture anchor
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Button Plates fixation system (Experimental): Patients receiving surgery fixed with Button Plates fixation system
  Interventions: Device: button plates fixation system
- Non-absorbable Suture Anchor (Active Comparator): Patients receiving surgery fixed with Non-absorbable suture anchor
  Interventions: Device: Non-absorbable Suture Anchor

INTERVENTIONS:
Device: button plates fixation system — The button plates fixation system consists of fixing plate, prefabricated mix, button and fuse. In the process of use, the fuse plays the role of guiding the fixed plate through, pulling the button and shortening the distance between the button and the fixed plate. The prefabricated mix is pre-worn between the button and the fixed plate, and the lead pulls the distance between the fixed plate and the button after tightening and fixing. Prefabricated mix, make mix tight and knot. Finish the preliminary work of fixing.
  Arms: Button Plates fixation system
Device: Non-absorbable Suture Anchor — A conventional device used in surgery for shoulder dislocation.
  Arms: Non-absorbable Suture Anchor

SUMMARY:
The purpose of this study is to conduct a comparative study through clinical trials to verify the safety and efficacy of the products in the experimental group for clinical use.

DETAILED DESCRIPTION:
The product of this clinical validation is the fixed button plate system, which is used for the reconstruction of the coracoclavicular ligament in the treatment of recurrent shoulder dislocation. The clinical trial was conducted to verify the rationality of its structural design, the convenience of its operation, and the effectiveness and safety of its clinical use. This trial was conducted in a parallel controlled trial design, the patients were divided into test and control groups to evaluate the safety and efficacy of the product.

ELIGIBILITY:
Inclusion Criteria:

1. a glenoid defect ≥10%
2. contact sport athletes with a glenoid defect < 10%
3. failure after Bankart repair.

Exclusion Criteria:

1. epilepsy
2. multidirectional shoulder instability
3. concomitant other lesions including rotator cuff tear, symptomatic acromioclavicular joint pathology or pathological involvement of the long head of the biceps
4. Follow-up was less than 2 years or incomplete follow-up data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Rowe score | before surgery
  The Rowe score is an internationally recognized scoring system for the assessment of shoulder function.
Rowe score | 3 months after surgery
  The Rowe score is an internationally recognized scoring system for the assessment of shoulder function.
Rowe score | 6 months after surgery
  The Rowe score is an internationally recognized scoring system for the assessment of shoulder function.

SECONDARY OUTCOMES:
ASES score | before surgery
  The American Shoulder and Elbow Surgeons (ASES) score is the most commonly used score to describe the function of patients' shoulder joints, ranging from 0 to 100. The higher the score, the better the function of patients' shoulder joints.
ASES score | 3 months after surgery
  The American Shoulder and Elbow Surgeons (ASES) score is the most commonly used score to describe the function of patients' shoulder joints, ranging from 0 to 100. The higher the score, the better the function of patients' shoulder joints.
ASES score | 6 months after surgery
  The American Shoulder and Elbow Surgeons (ASES) score is the most commonly used score to describe the function of patients' shoulder joints, ranging from 0 to 100. The higher the score, the better the function of patients' shoulder joints.

CONTACTS AND LOCATIONS:
Overall Officials: Guoqing Cui, Study Chair — Peking University Third Hospital
Locations (1):
- PekingUTH, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No